CLINICAL TRIAL: NCT07043946
Title: A Phase 1b/2a, Open-Label, Sequential-Cohort, Dose Escalation and Expansion Study to Evaluate Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, and Preliminary Clinical Effectiveness of Budoprutug (TNT119) in Subjects With Immune Thrombocytopenia (ITP)
Brief Title: A Phase 1b/2a Study of Budoprutug in Subjects With Immune Thrombocytopenia (ITP)
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Climb Bio, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: TNT119-ITP-201
Record Dates: First submitted 2025-06-20; First posted 2025-06-29 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Immune Thrombocytopenia (ITP); ITP; Biologics; Monoclonal; Anti-CD19
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic

STUDY DESIGN:
Intervention Model Description: This is an open-label study in which subjects will be enrolled into three dose ascending cohorts. Each subject's participation will last approximately 51 weeks including the Screening and Qualifying Visits (up to 3 weeks), Treatment Period (2 weeks), and follow-up visits though Week 48. Following completion of the dose escalation phase, additional subjects will be enrolled into an expansion cohort at the selected dose level(s) identified in Part 1b.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Cohort 1: Dose Level A (Experimental): Single IV dose of study product on Day 1 and on Day 15
  Interventions: Drug: Budoprutug
- Cohort 2: Dose Level B (Experimental): Single IV dose of study product on Day 1 and on Day 15
  Interventions: Drug: Budoprutug
- Cohort 3: Dose Level C (Experimental): Single IV dose of study product on Day 1 and on Day 15
  Interventions: Drug: Budoprutug
- Dose Expansion Cohort (Experimental): Single IV dose of study product on Day 1 and Day 15
  Interventions: Drug: Budoprutug

INTERVENTIONS:
Drug: Budoprutug — Single IV dose of study product on Day 1 and Day 15
  Other Names: TNT119

SUMMARY:
The main objective is to assess the safety and tolerability of budoprutug in adults with ITP. Pharmacokinetics, pharmacodynamics, and preliminary clinical efficacy will also be assessed.

DETAILED DESCRIPTION:
Budoprutug is a humanized, immunoglobulin (Ig) G1 monoclonal antibody that selectively binds to CD19 and is projected to deplete targeted cells through antibody-dependent cellular cytotoxicity. This Phase 1b/2a, open-label, sequential-cohort, dose escalation and expansion study will evaluate the safety, tolerability, PK, PD, and preliminary clinical effectiveness of budoprutug in subjects with ITP. Budoprutug will be administered as two (2) IV infusions 14 days apart in ascending dose cohorts of patients aged 18 years and above with a platelet count < 30,000/µL despite an adequate trial of at least one prior therapeutic attempt.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 years at the time of consent.
2. Platelet count < 30,000/µL despite an adequate trial of at least one prior therapeutic attempt. Platelet counts of < 30,000/µL must be confirmed on 2 occasions at least 5 days apart, but no more than 14 days apart.
3. Partial thromboplastin time < 1.5 x upper limit of normal (ULN), prothrombin time < 1.5 x ULN, total bilirubin < 1.5 x ULN unless due to Gilbert's syndrome, or an international normalized ratio < 1.5 at screening.

Exclusion Criteria:

1. CD19+ B cell count < 80 cells/µL at Screening, or < 40 cells/µL if B-cell depleting therapy was received within 24 weeks to 2 years prior.
2. Diagnosis of paroxysmal nocturnal hemoglobinuria, Evan's Syndrome, or other bleeding disorders affecting safety or data integrity.
3. Prior B-cell depleting therapy (e.g., rituximab) within 24 weeks before first dose or planned during the study.
4. Chronic use of anticoagulants or antiplatelet agents (e.g., aspirin, NSAIDs, thienopyridines) within 14 days before dosing through follow-up. Intermittent NSAID use is allowed.
5. Immunosuppressants (excluding corticosteroids) within 30 days or 5× half-life before Screening; alkylating agents within 180 days.
6. IVIg treatment within 90 days prior to Screening.
7. Active ITP treatment (other than steroids or TPO agonists) within 30 days or 5× half-life before first dose, unless approved by Medical Monitor.
8. Active, chronic, or latent infections including hepatitis B/C or HIV.
9. Active TB or high TB risk.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-06-30 (Actual); Primary Completion 2027-08 (Estimated); Study Completion 2028-08 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events (TEAEs) | Up to week 48
  Number of participants experiencing TEAEs, graded per NCI CTCAE v5.0.

SECONDARY OUTCOMES:
Area Under the Curve (AUC) | Up to week 48
  Measurement of the area under the drug concentration-time curve.
Maximum Observed Plasma Concentration (Cmax) | Up to week 48
  Measurement of the maximum observed plasma concentration.
Time to Maximum Observed Concentration (Tmax) | Up to week 48
  Measurement of the time to maximum observed concentration.
Terminal Half-Life (T1/2) | Up to week 48
  Measurement of the terminal half-life in days.
Apparent Clearance (CL/F) | Up to week 48
  Measurement of the apparent clearance in L/hour.
Change from Baseline in CD20+ B-cell Count | Up to week 48
  Change in absolute peripheral CD20+ B-cell count
Change in Platelet Count | Up to week 48
  Change in platelet count over time
Proportion of Participants with stable, partial or complete platelet response | Up to week 48
  Percentage of participants with stable, partial or complete platelet response.
Incidence of Anti-Drug Antibodies (ADAs) | Up to week 48
  Number of participants with detectable ADAs.
Steroid Discontinuation Rate | Up to week 48
  % of baseline steroid users who discontinue steroids.

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Climb Bio, Inc.
Locations (19):
- Bulgaria (3):
  - Climb Bio Investigative Site #359202, Plovdiv
  - Climb Bio Investigative Site #359203, Plovdiv
  - Climb Bio Investigative Site #359201, Sofia
- Greece (4):
  - Climb Bio Investigative Site #300204, Athens, Attica
  - Climb Bio Investigative Site #300203, Chaïdári, Attica
  - Climb Bio Investigative Site #300202, Ioannina
  - Climb Bio Investigative Site #300201, Thessaloniki
- Serbia (3):
  - Climb Bio Investigative Site #381201, Belgrade
  - Climb Bio Investigative Site #381202, Belgrade
  - Climb Bio Investigative Site #381203, Novi Sad
- Spain (4):
  - Climb Bio Investigative Site #340206, Burgos
  - Climb Bio Investigative Site #340204, Madrid
  - Climb Bio Investigative Site #340202, San Pedro
  - Climb Bio Investigative Site #340203, Valencia
- Ukraine (5):
  - Climb Investigative Site #380204, Ivano-Frankivsk
  - Climb Investigative Site #2380203, Kyiv
  - Climb Investigative Site #380202, Kyiv
  - Climb Investigative Site #380206, Kyiv
  - Climb Investigative Site #380201, Lviv

IPD SHARING:
Plan to Share IPD: No